CLINICAL TRIAL: NCT05514886
Title: Evaluation of Molecular Point-of-care Xpert® Xpress SARS-CoV-2 Detection Implementation in Resource-limited Settings
Acronym: EXPERT-CoV-2
Status: Completed | Type: Observational
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: University of Kinshasa (Other); Research Institute for Health Sciences - Burkina Faso (Unknown); Universiteit Antwerpen, Belgium (Unknown); Københavns Universitet (Other); Universidad de Valencia, Spain (Unknown)
Responsible Party: Principal Investigator, Daniel T Minja, PhD, Principal Investigator, National Institute for Medical Research, Tanzania
Other Study IDs: EXPERT-CoV-2
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Surgical Instruments

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasopharyngeal or nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Gene Expert molecular Point-of-Care (POC) (Xpert® Xpress SARS-CoV-2/Flu/RSV test — POC viral load (VL) assay in improving the availability of SARS-CoV-2 detection for COVID-19 patient management in decentralized healthcare facilities of resource-constrained settings in Tanzania, DR Congo and Burkina Faso.

SUMMARY:
This study evaluated the diagnostic accuracy and effectiveness of POC viral load (VL) assay in improving the availability of SARS-CoV-2 detection for COVID-19 patient management in decentralised healthcare facilities of resource-constrained settings in Tanzania, DR Congo and Burkina Faso.

DETAILED DESCRIPTION:
Project Title: Evaluation of molecular point-of-care Xpert® Xpress SARS-CoV-2 detection implementation in resource limited settings (RIA2020EF-2990) - EXPERT-CoV-2

Clinical Trial Registration: NCT05514886

Principal Investigator: Dr Daniel T. R Minja, NIMR- Tanga Centre, Korogwe Research Station, Tanzania

Collaborating Partners: University of Kinshasa, DR Congo, Research Institute for Health Sciences, Burkina Faso, University of Copenhagen, Denmark, University of Antwerp, Belgium, University of Valencia, Spain

Funding: This project (RIA2020EF-2990) is part of the EDCTP2 programme supported by the European Union.

Date: 17th July 2024

Background: Rapid diagnostic tests of individuals infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) are the cornerstone to implementing early case detection and management to control the spread of the deadly virus. RT-PCR is the gold standard for the detection of SARS-CoV-2 but its availability and usability is impeded by fragmented laboratory infrastructure in LMICs and even when available it's only found in reference labs.

The recent development of the Gene Expert molecular Point-of-Care (POC) (Xpert® Xpress SARS-CoV-2/Flu/RSV test, Cepheid Sunnyvale, CA) for SARS-CoV-2 testing in the clinics with results delivery within hours of sample collection has been vital in resolving the turnaround time (TAT). GeneXpert has been widely rolled out within national tuberculosis (TB) and HIV programmes across Africa. However, evaluation of its diagnostic accuracy and the feasibility of its integration into the TB/HIV programme has not been evaluated in resource-constrained settings.

Study objective: This study is envisaged to evaluate the diagnostic accuracy and effectiveness of POC viral load (VL) assay in improving the availability of SARS-CoV-2 detection for COVID-19 patient management in decentralised healthcare facilities of resource-constrained settings in Tanzania, DR Congo and Burkina Faso.

Methods and Results: This study was conducted in Tanzania, Burkina Faso and DR Congo between 21st July 2021 and February 2024. Data analyses are ongoing and further updates will be made available once the final phylogenetic analyses are completed and ready for publication, details of the clades and variants will also be available.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years and above presenting with symptoms as indicated in national COVID-19 standard cases definitions or
* Presence of one or more respiratory symptoms (fever (defined as >37.5°C), Persistent coughs, headache, myalgia, sore throat ) or One risk factor for COVID-19, including known contact with a patient with COVID-19, underlying comorbidities, smoking.
* Provision of an informed consent/assent (for minors aged 11-17 years) by themselves or parents/guardians to participate

Exclusion Criteria:

* Inability or unwillingness to give written informed consent/assent.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals age 5 years and above with respiratory symptoms suggestive of SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 3429 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with SARS-CoV-2 infection | 24 months
  The study will screen patients with respiratory tract infections suggestive of SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: DANIEL TR MINJA, PhD, Principal Investigator — National Institute for Medical Research, Tanzania
Locations (1):
- Nimr Korogwe, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided
This will be discussed in the consortium and once consensus has been reached, it will be decided on which information and data will be shared.